CLINICAL TRIAL: NCT03239353
Title: A Phase 1, Randomized, Partially-Blind, Parallel-Group, Active and Placebo Controlled Study to Evaluate the Safety and Pharmacokinetics of Single Oral Doses of Entecavir Extended Release (XR) in Healthy Subjects
Brief Title: A Phase 1 Study to Evaluate the Safety and Pharmacokinetics of Entecavir Extended Release (XR) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aucta Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UAP008C001
Record Dates: First submitted 2017-07-27; First posted 2017-08-04 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: HBV
MeSH Terms: interventions — entecavir

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- 1.5 mg ETV XR tablet (Active Comparator)
  Interventions: Drug: Entecavir
- 3 mg ETV XR tablet (Active Comparator)
  Interventions: Drug: Entecavir
- 6 mg ETV XR tablet (Active Comparator)
  Interventions: Drug: Entecavir
- Placebo-to-match 1.5 mg ETV XR tablet (Placebo Comparator)
  Interventions: Drug: Entecavir
- 0.5 mg ETV IR tablet (Other)
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Entecavir — Study drug (entecavir or placebo) will be administered with 240 mL of water following an overnight fast (no food or drink, except water, for at least 10 hours). Subjects will be required to fast (no food or beverages other than water) until after collection of the 4-hour blood draw.
  Other Names: placebo

SUMMARY:
This is a phase 1, randomized, parallel-group, single-center study in healthy adult subjects. The study will be conducted in two parts sequentially:

Part 1 is an open-label, two-arm, active-controlled design to evaluate the PK and safety of single oral dose of ETV XR tablet (1.5 mg) in healthy subjects. Part 1 will consist of 16 healthy subjects.

Part 2 is a double-blind, three-arm, placebo-controlled design to evaluate the PK and safety of higher oral doses of ETV XR tablet (3 mg and 6 mg) in healthy subjects. Part 2 will consist of 24 healthy subjects.

ELIGIBILITY:
Inclusion criteria:

Subjects will be considered for enrollment in the study if they meet all of the inclusion criteria and none of the exclusion criteria.

1. Male or female aged between 18 and 55 years (inclusive). Body weight ≥ 50 kg for males, and ≥45 kg for females and Body Mass Index (BMI) between 18 and 28 kg/m2 (inclusive), BMI(kg/m2) = body weight(kg)/{height(m)}2;
2. Ability to fully understand the purpose, characteristic, method and the possible adverse effects of the trial, and voluntarily signed Informed Consent obtained before any trial-related procedures are performed;
3. Ability to comply with the requirements of this trial protocol, including refrain from strenuous exercise/activity 3 days prior to Day -1 (admission) and for 3 days prior to the Day 8, Day 15 and the final follow-up visit on Day 22through the duration of the study
4. Have a creatinine clearance (CLCr) ≥ 80 mL/min;
5. Male subjects and female subjects of child bearing potential must be willing to practice effective contraception during the study and been willing and able to continue contraception for 90 days after their dose of the study treatment;
6. Male subjects must refrain from sperm donation from Day -1 through completion of the study and continuing for at least 90 days from the date of last dose of study drug;
7. Subjects must refrain from blood donation from Screening through completion of the study and continuing for at least 30 days from date of last dose of study drug;
8. AST, ALT and bilirubin ≤ 1.5xULN (isolated bilirubin > 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%);
9. Must, in the opinion of the Investigator, be in good health based upon medical history, physical examination (including vital signs), and screening laboratory evaluations (hematology, chemistry, and urinalysis must fall within the normal range of the central laboratory reference ranges unless the results have been determined by the Investigator to have no clinical significance).

Exclusion criteria:

A subject meeting any of the following criteria will be excluded from the study:

1. Current or a history of any clinically significant medical illness or medical disorders the investigator considers should exclude including (but not limited to) neurological disease, cardiovascular disease, hepatic or renal disease, gastrointestinal tract disease (such as dysphagia, gastrointestinal ulcers), respiratory disease, metabolism, skeletal system diseases or other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs;
2. Has a positive result from serology examination for hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV);
3. There are drug-dependent or drug abuse history, or urine drug abuse screening positive;
4. Subject smoked more than 5 cigarettes or other tobacco or nicotine-containing products within 1 month prior to dosing and is unwilling to abstain from smoking for 48 hours prior to check-in (Day -1)ing, for the duration of the confinement period and at each follow-up visit;
5. Has used an alcohol consumption of more than 14 units of alcohol per week (1 unit of alcohol is equivalent to 360 mL of beer or 45 mL of spirits with 40 % of alcohol or 150 mL of wine) within 6 months prior to screening or taking products containing alcohol 48 hours prior to IMP administration;
6. Participated in any drug or medical device clinical trial within 3 months prior to screening;
7. Pregnant or breastfeeding women or pregnancy testing is positive;
8. Have taken any prescription medications, over-the-counter medications, supplements or herbal products within 14 days, or 5 half-lives (whichever is longer), of study drug dosing, with the exception of paracetamol and hormonal contraceptive medications, unless in the opinion of the Investigator and/or Medical Monitor that the substance would not have any material impact on participant safety or the quality of study data;
9. Donated blood greater than 400 mL or significant blood loss equivalent to 400 mL or received blood transfusion within 3 months of screening; Or donated blood greater than 200 ml or significant blood loss equivalent to 200 mL within 1 months prior to screening;
10. Has infectious diseases within four weeks at screening (in the opinion of the investigator would pose a risk for participation in this study), severe trauma, or a history of major surgery within 3 months;
11. Cannot tolerate venepuncture or cannulation;
12. Consumption of grapefruit, grapefruit juice, cranberries, or products containing Seville oranges (fruit juices, marmalade, jam, etc) within 7 days prior to study drug dosing; consumption of caffeine-containing products within 48 hours of study drug dosing;
13. Have been vaccinated within 90 days of study dosing, with the exception of licensed intranasal or intramuscular influenza vaccine ≤ 14 days prior to dosing.
14. Have severe multiple allergies and / or severe allergies (including latex / heparin allergy) history, or has hypersensitivity or significant intolerance to prescription drugs or over-the-counter drugs or food;
15. Subjects who, in the opinion of the Investigator, should not participate in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
To characterize the Pharmacokinetics (PK) of ETV XR tablet after single oral doses in healthy subjects. | 22 days
  Peak Plasma Concentration(Cmax)
To characterize the Pharmacokinetics (PK) of ETV XR tablet after single oral doses | 22 days
  Area under the plasma concentration versus time curve (AUC)
To characterize the Pharmacokinetics (PK) of ETV XR tablet after single oral doses | 22 days
  peak time (Tmax)
To characterize the Pharmacokinetics (PK) of ETV XR tablet after single oral doses | 22 days
  Relative bioavailability (Frelative)
To characterize the Pharmacokinetics (PK) of ETV XR tablet after single oral doses | 22 days
  half life (t1/2)

SECONDARY OUTCOMES:
To assess ETV XR tablet in healthy subjects. | 22 days
  adverse events
To assess ETV XR tablet in healthy subjects. | 22 day
  laboratory abnormalities
To assess ETV XR tablet in healthy subjects. | 22 days
  vital signs
To assess ETV XR tablet in healthy subjects. | 22 days
  12-lead electrocardiograms (ECGs)
To evaluate the dose linearity of ETV XR tablet | 60 days
  1.5mg, 3mg and 6mg PK linearity

CONTACTS AND LOCATIONS:
Locations (1):
- Linear Clinical Research Ltd, Nedlands, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No